CLINICAL TRIAL: NCT04740905
Title: A Phase III, Multicenter, Randomized, Double-Masked, Active Comparator-Controlled Study to Evaluate the Efficacy and Safety of Faricimab in Patients With Macular Edema Secondary to Branch Retinal Vein Occlusion
Brief Title: A Study to Evaluate the Efficacy and Safety of Faricimab in Participants With Macular Edema Secondary to Branch Retinal Vein Occlusion
Acronym: BALATON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR41984; 2020-000440-63 (EudraCT Number)
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Macular Edema; Branch Retinal Vein Occlusion
Keywords: BRVO
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — faricimab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) (Experimental): In Part 1 (Day 1 through Week 24), participants randomly assigned to Arm A will receive faricimab 6 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections). In Part 2 (from Week 24 to Week 72), participants will receive faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure will be administered during study visits at which no faricimab treatment is administered (according to the PTI dosing regimen).
  Interventions: Drug: Faricimab; Procedure: Sham Procedure
- Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2) (Active Comparator): In Part 1 (Day 1 through Week 24), participants randomly assigned to Arm B will receive aflibercept 2 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections). In Part 2 (from Week 24 to Week 72), participants will receive faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure will be administered during study visits at which no faricimab treatment is administered (according to the PTI dosing regimen).
  Interventions: Drug: Faricimab; Drug: Aflibercept; Procedure: Sham Procedure

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered by intravitreal (IVT) injection as specified in each treatment arm.
  Other Names: VABYSMO®; faricimab-svoa; RO6867461; RG7716
Drug: Aflibercept — Aflibercept 2 mg will be administered by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections).
  Other Names: Eylea
  Arms: Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Procedure: Sham Procedure — The sham is a procedure that mimics an intravitreal (IVT) injection, but involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.

SUMMARY:
This is a Phase III, multicenter, randomized, double-masked, active comparator-controlled, parallel-group study evaluating the efficacy, safety, and pharmacokinetics of faricimab administered by intravitreal (IVT) injection at 4-week intervals until Week 24, followed by a double-masked period of study without active control to evaluate faricimab administered according to a personalized treatment interval (PTI) dosing regimen in participants with macular edema due to branch retinal vein occlusion (BRVO).

ELIGIBILITY:
Inclusion Criteria:

* Foveal center-involved macular edema due to branch retinal vein occlusion (BRVO), diagnosed no longer than 4 months prior to the screening visit
* Best-corrected visual acuity (BCVA) of 73 to 19 letters, inclusive (20/40 to 20/400 approximate Snellen equivalent) on Day 1
* Sufficiently clear ocular media and adequate pupillary dilatation to allow acquisition of good quality retinal images to confirm diagnosis
* For women of childbearing potential: agreement to remain abstinent or use contraception, and agreement to refrain from donating eggs during the treatment period and for 3 months after the final dose of study treatment

Exclusion Criteria:

* Any major illness or major surgical procedure within 1 month before screening
* Uncontrolled blood pressure
* Stroke (cerebral vascular accident) or myocardial infarction within 6 months prior to Day 1
* Pregnant or breastfeeding, or intending to become pregnant during the study

Ocular Exclusion Criteria for Study Eye:

* History of previous episodes of macular edema due to RVO or persistent macular edema due to RVO diagnosed more than 4 months before screening
* Any current ocular condition which, in the opinion of the investigator, is currently causing or could be expected to contribute to irreversible vision loss due to a cause other than macular edema due to RVO in the study eye (e.g., ischemic maculopathy, Irvine-Gass syndrome, foveal atrophy, foveal fibrosis, pigment abnormalities, dense subfoveal hard exudates, or other non-retinal conditions)
* Macular laser (focal/grid) in the study eye at any time prior to Day 1
* Panretinal photocoagulation in the study eye within 3 months prior to Day 1 or anticipated within 3 months of study start on Day 1
* Any prior or current treatment for macular edema; macular neovascularization, including diabetic macular edema (DME) and neovascular age-related macular degeneration (nAMD); and vitreomacular-interface abnormalities, including, but not restricted to, IVT treatment with anti-VEGF, steroids, tissue plasminogen activator, ocriplasmin, C3F8, air or periocular injection
* Any prior intervention with verteporfin photodynamic therapy, diode laser, transpupillary thermotherapy, or vitreo-retinal surgery including sheatotomy
* Any prior steroid implant use including dexamethasone intravitreal implant (Ozurdex) and fluocinolone acetonide intravitreal implant (Iluvien)

Ocular Exclusion Criteria for Both Eyes:

* Prior IVT administration of faricimab in either eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Active periocular, ocular or intraocular inflammation or infection (including suspected) in either eye on Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (150):
- United States (39):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - California Eye Specialists Medical group Inc., Pasadena, California
  - Retina Consultants, San Diego, Poway, California
  - Retina Consultants of Southern Colorado PC, Colorado Springs, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Florida Eye Associates, Melbourne, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Prairie Retina Center, Springfield, Illinois
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - Tufts Medical Center; Ophthalmology, Boston, Massachusetts
  - Assoc Retinal Consultants PC, Royal Oak, Michigan
  - VitreoRetinal Surgery, PLLC.; DBA Retina Consultants of Minnesota, Edina, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Retina Associates of NJ, Teaneck, New Jersey
  - Long Is. Vitreoretinal Consult, Hauppauge, New York
  - Retina Vit Surgeons/Central NY, Liverpool, New York
  - Graystone Eye, Hickory, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina & Vitreous of Texas, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, PLLC, Salt Lake City, Utah
- Argentina (9):
  - Fundacion Zambrano, CABA
  - Centro Oftalmológico Dr. Charles S.A., Capital Federal
  - Oftalmos, Capital Federal
  - Hospital Italiano; Ophtalmology, Capital Federal
  - Buenos Aires Mácula, Ciudad Autonoma Buenos Aires
  - Oftar, Mendoza
  - Centro Oftalmólogos Especialistas, Rosario
  - Grupo Laser Vision, Rosario
  - Organizacion Medica de Investigacion, San Nicolás
- Australia (6):
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Save Sight Institute, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- LKH-Univ.Klinikum Graz; Universitäts-Augenklinik, Graz, Austria
- Brazil (4):
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Botelho Hospital da Visao, Blumenau, Santa Catarina
  - Universidade Federal de Sao Paulo - UNIFESP*X; Oftalmologia, São Paulo, São Paulo
  - Hosp de Olhos de Sorocaba, Sorocaba, São Paulo
- China (14):
  - Beijing Hospital of Ministry of Health, Beijing
  - The Second Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin
  - The Affiliated Eye Hospital of Nanjing Medical University, Nanjing
  - Shanghai Tenth People's Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - He Eye Specialist Shenyang Hospital, Shenyang
  - Tianjin Eye Hospital, Tianjin
  - Tianjin Medical University Eye Hospital, Tianjin
  - Eye Hospital, Wenzhou Medical University, Wenzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - Henan Provincial Eye Hosptial, Zhengzhou
- Czechia (4):
  - Faculty Hospital Ostrava; Ophthalmology clinic, Ostrava
  - Faculty Hospital Kralovske Vinohrady; Ophthalmology clinic, Prague
  - AXON Clinical, Prague
  - Nemocnice Sokolov, Sokolov
- France (2):
  - Chi De Creteil; Ophtalmologie, Créteil
  - Hopital Lariboisiere; Ophtalmologie, Paris
- Germany (3):
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Universitätsmedizin Göttingen Georg-August-Universität; Klinik für Augenheilkunde, Göttingen
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH; Augenklinik, Ludwigshafen
- Hong Kong (2):
  - Queen Mary Hospital; Department of Ophthalmology, Hong Kong
  - Hong Kong Eye Hospital; CUHK Eye Centre, Mong Kok
- Hungary (4):
  - Budapest Retina Associates Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont; Szemeszeti Klinika, Debrecen
  - Ganglion Medial Center, Pécs
  - Szegedi Tudományegyetem ÁOK; Department of Ophtalmology, Szeged
- Israel (5):
  - Rambam Medical Center; Opthalmology, Haifa
  - Hadassah MC; Ophtalmology, Jerusalem
  - Rabin MC; Ophtalmology, Petah Tikva
  - Kaplan Medical Center; Ophtalmology, Rehovot
  - Tel Aviv Sourasky MC; Ophtalmology, Tel Aviv
- Italy (3):
  - Fondazione Ptv Policlinico Tor Vergata Di Roma;U.O.S.D. Patologie Renitiche, Rome, Lazio
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena;U.O.C Oculistica, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria Careggi; S.O.D. Oculistica, Florence, Tuscany
- Japan (15):
  - Sugita Eye Hospital, Aichi
  - Nagoya University Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - Aichi Medical University Hospital, Aichi
  - Toho University Sakura Medical Center, Chiba
  - Hayashi Eye Hospital, Fukuoka
  - Southern TOHOKU Eye Clinic, Fukushima
  - Asahikawa Medical University Hospital, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center (Hyogo AGMC), Hyōgo
  - Hyogo Medical University Hospital, Hyōgo
  - Kozawa eye hospital and diabetes center, Ibaraki
  - Kyoto University Hospital, Kyoto
  - Tokushima University Hospital, Tokushima
  - Nihon University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
- Poland (10):
  - Specjalistyczny O?rodek Okulistyczny Oculomedica, Bydgoszcz
  - Szpital Specjalistyczny nr 1; Oddzial Okulistyki, Bytom
  - Dobry Wzrok Sp Z O O, Gda?sk
  - Poradnia Okulistyczna i Salon Optyczny w Gliwicach- PRYZMAT, Gliwice
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - Centrum Medyczne Dietla 19 Sp. Z O.O., Krakow
  - Centrum Medyczne Pulawska SP. z o.o., Piaseczno
  - Lens Clinic, Rybnik
  - Caminomed, Tarnowskie Góry
  - Centrum Zdrowia MDM, Warsaw
- Portugal (3):
  - Centro Hospitalar E Universitário de Coimbra EPE - Serviço Oftalmologia; Serviço Oftalmologia, Coimbra
  - Espaco Medico Coimbra, Coimbra
  - Centro Hospitalar Universitário do Porto ? Hospital de Santo António; Servico de Oftalmologia, Porto
- Russia (3):
  - Clinic Optimed, Ufa, Bashkortostan Republic
  - Clinics of Eye Diseases, LLC, Kazan', Tatarstan Republic
  - ?Intersec. Research and Technology Complex ?Eye Microsurgery? n a Fyodorov Irkutsk branch, Irkutsk
- Singapore (2):
  - Singapore Eye Research Institute, Singapore
  - Tan Tock Seng Hospital; Ophthalmology Department, Singapore
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Clinica Universitaria de Navarra; Servicio de Oftalmologia, Pamplona, Navarre
  - Oftalvist Valencia, Burjassot, Valencia
  - Hospital dos de maig; servicio de oftalmologia, Barcelona
  - Clinica Baviera; Servicio Oftalmologia, Madrid
  - Hospital Universitario Rio Hortega; Servicio de Oftalmologia, Valladolid
- Taiwan (4):
  - Changhua Christian Hospital; Department of Ophthalmology, Changhua
  - Taipei Veterans General Hospital; Ophthalmology, Taipei
  - Chang Gung Medical Foundation - Linkou; Ophthalmology, Taoyuan District
  - National Taiwan University Hospital; Ophthalmology, Zhongzheng Dist.
- United Kingdom (6):
  - Belfast Health and Social Care Trust, ROYAL VICTORIA HOSPITAL, Belfast
  - Bristol Eye Hospital;Retinal Treatment and Research Unit, Bristol
  - University Hospital of Wales, Cardiff
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - St James University Hospital, Leeds
  - Central Middlesex Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Romano F, Lamanna F, Gabrielle PH, Teo KYC, Battaglia Parodi M, Iacono P, Fraser-Bell S, Cornish EE, Nassisi M, Viola F, Agarwal A, Samanta A, Chhablani J, Staurenghi G, Invernizzi A. Update on Retinal Vein Occlusion. Asia Pac J Ophthalmol (Phila). 2023 Mar-Apr 01;12(2):196-210. doi: 10.1097/APO.0000000000000598. Epub 2023 Feb 14. PMID 36912792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 768 patients were screened; 9 of these patients were rescreened and randomized in the study. A total of 215 patients failed screening due to not meeting the inclusion criteria. A total of 553 patients with BRVO were randomized 1:1 into the study: 276 to the faricimab Q4W arm and 277 to the aflibercept Q4W arm.
Groups:
- Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2): In Part 1 (Day 1 through Week 24), participants were randomly assigned to Arm A to receive faricimab 6 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections). In Part 2 (from Week 24 to Week 72), participants received faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure was administered during study visits at which no faricimab treatment was administered (according to the PTI dosing regimen).
- Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2): In Part 1 (Day 1 through Week 24), participants were randomly assigned to Arm B to receive aflibercept 2 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections). In Part 2 (from Week 24 to Week 72), participants received faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure was to be administered during study visits at which no faricimab treatment was administered (according to the PTI dosing regimen).
Period: Part 1 (Baseline up to Week 24)
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Started (Intent-to-Treat (ITT) Population) | 276 (All randomized participants) | 277 (All randomized participants)
Received at Least One Dose of Study Drug (Safety-Evaluable Population) | 276 | 274
Completed (Completed Part 1) | 271 | 274
Not Completed | 5 | 3
Not completed — Protocol Violation | 0 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0
Period: Part 2 (Week 24 to Week 72)
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Started | 271 | 274
Completed | 245 | 244
Not Completed | 26 | 30
Not completed — Withdrawal by Subject | 13 | 12
Not completed — Lost to Follow-up | 7 | 6
Not completed — Adverse Event | 0 | 4
Not completed — Physician Decision | 0 | 4
Not completed — Patient Missed Week 72 Visit Due to SAE | 1 | 1
Not completed — Death | 1 | 2
Not completed — Non-Compliance With Study Drug | 2 | 1
Not completed — Patient Could Not Return to Hospital Due to COVID-19 Epidemic | 1 | 0
Not completed — Patient Refused to Continue Study | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population: All global participants who were randomized in the study, according to the assigned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2) | Total
Number analyzed (Participants) | 276 | 277 | 553
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (10.7) | 63.8 (10.6) | 64.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 147 | 280
  Male | 143 | 130 | 273
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 51 | 98
  Not Hispanic or Latino | 224 | 224 | 448
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 90 | 94 | 184
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 7 | 13
  White | 172 | 172 | 344
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Rest of the World | 129 | 128 | 257
  Asia | 85 | 85 | 170
  USA and Canada | 62 | 64 | 126
Number of Participants by the Eye (Left or Right) Chosen as the Study Eye [Count of Participants; unit: Participants]
  Left Eye | 140 | 127 | 267
  Right Eye | 136 | 150 | 286
Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye [Mean (Standard Deviation); unit: ETDRS Letters] | 57.50 (13.04) | 57.64 (12.15) | 57.57 (12.59)
Number of Participants by the BCVA Letter Score Categories in the Study Eye [Count of Participants; unit: Participants]
  ≤54 Letters (20/80 or Worse) | 89 | 90 | 179
  ≥55 Letters (20/80 or Better) | 187 | 187 | 374

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye at Week 24
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. The Mixed Model of Repeated Measures (MMRM) analysis included the categorical covariates of treatment arm, visit, visit-by-treatment arm interaction, baseline BCVA (continuous), and randomization stratification factors [baseline BCVA (≥55 and ≤54 letters), and region (U.S. and Canada, Asia, and rest of the world)] as fixed effects. An unstructured covariance structure was used. Missing data were implicitly imputed by MMRM model assuming missing at random. Treatment policy strategy (i.e., all observed values used) was applied to all intercurrent events (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). 95% CI is a rounding of 95.03% CI.
Time Frame: From Baseline through Week 24
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Groups:
- Arm A: Faricimab Q4W (Part 1): In Part 1 (Day 1 through Week 24), participants randomly assigned to Arm A were to receive faricimab 6 milligrams (mg) administered by intravitreal (IVT) injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections).
- Arm B: Aflibercept Q4W (Part 1): In Part 1 (Day 1 through Week 24), participants randomly assigned to Arm B were to receive aflibercept 2 milligrams (mg) administered by intravitreal (IVT) injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections).
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
ETDRS Letters | 16.9 [15.7 to 18.1] | 17.5 [16.3 to 18.6]
Statistical Analysis 1: Comparison: Arm A: Faricimab Q4W (Part 1) vs Arm B: Aflibercept Q4W (Part 1); The null hypothesis, H0: μ(faricimab) - μ(aflibercept) ≤-4 letters; the alternative hypothesis, Ha: μ(faricimab) - μ(aflibercept) >-4 letters. The final sample size provided >90% power for the non-inferiority assessment (at a one-sided 0.02485 significance level); Test type: Non-Inferiority — If the lower bound of a two-sided 95% confidence interval (CI) for the difference in adjusted means of the two treatments (faricimab minus aflibercept) is greater than -4 letters (the non-inferiority margin), then faricimab is considered non-inferior to aflibercept; Difference in Adjusted Means = -0.6, 95% CI 2-sided [-2.2 to 1.1], Standard Error of Mean 0.84 — The treatment difference in adjusted means of change from baseline BCVA is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept. MMRM adjustments are listed in the outcome measure description
Statistical Analysis 2: Comparison: Arm A: Faricimab Q4W (Part 1) vs Arm B: Aflibercept Q4W (Part 1); The final sample size provided >80% power for a 3.5-letter superiority assessment of faricimab over aflibercept; Test type: Superiority; p = 0.4978, Mixed Model of Repeated Measures — Tested at a two-sided 0.0497 significance level; Difference in Adjusted Means = -0.6, 95% CI 2-sided [-2.2 to 1.1], Standard Error of Mean 0.84 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Part 1: Change From Baseline in BCVA in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
ETDRS Letters
  Week 4 | 11.5 [10.5 to 12.5] | 12.4 [11.4 to 13.4]
  Week 8 | 13.7 [12.6 to 14.7] | 15.1 [14.1 to 16.2]
  Week 12 | 15.1 [14.0 to 16.2] | 15.9 [14.8 to 17.0]
  Week 16 | 15.5 [14.4 to 16.6] | 16.5 [15.4 to 17.7]
  Week 20 | 16.3 [15.2 to 17.4] | 17.3 [16.1 to 18.4]
  Week 24 | 16.9 [15.7 to 18.1] | 17.5 [16.3 to 18.6]

3. Secondary Outcome: Part 1: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye at Week 24
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≥55 and ≤54 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants | 56.1 [50.4 to 61.9] | 60.4 [54.7 to 66.0]
Statistical Analysis 1: Comparison: Arm A: Faricimab Q4W (Part 1) vs Arm B: Aflibercept Q4W (Part 1); Test type: Other; Difference in CMH Weighted Percentage = -4.3, 95% CI 2-sided [-12.3 to 3.8]

4. Secondary Outcome: Part 1: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 34.3 [28.9 to 39.8] | 36.9 [31.5 to 42.3]
  Week 8 | 41.2 [35.6 to 46.9] | 46.7 [41.0 to 52.3]
  Week 12 | 51.0 [45.3 to 56.7] | 52.1 [46.3 to 57.8]
  Week 16 | 53.6 [47.8 to 59.3] | 56.4 [50.8 to 62.1]
  Week 20 | 56.1 [50.3 to 61.8] | 58.9 [53.3 to 64.6]
  Week 24 | 56.1 [50.4 to 61.9] | 60.4 [54.7 to 66.0]

5. Secondary Outcome: Part 1: Percentage of Participants Gaining ≥10 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 57.5 [51.8 to 63.3] | 59.2 [53.6 to 64.9]
  Week 8 | 69.1 [63.8 to 74.5] | 69.0 [63.6 to 74.4]
  Week 12 | 75.0 [69.9 to 80.1] | 74.8 [69.7 to 79.8]
  Week 16 | 72.1 [66.9 to 77.3] | 76.6 [71.6 to 81.5]
  Week 20 | 75.3 [70.3 to 80.4] | 79.1 [74.3 to 83.9]
  Week 24 | 77.5 [72.6 to 82.4] | 77.3 [72.4 to 82.2]

6. Secondary Outcome: Part 1: Percentage of Participants Gaining ≥5 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 75.7 [70.7 to 80.7] | 79.1 [74.4 to 83.9]
  Week 8 | 84.0 [79.7 to 88.3] | 88.1 [84.3 to 91.9]
  Week 12 | 87.0 [83.1 to 90.9] | 87.0 [83.1 to 91.0]
  Week 16 | 85.9 [81.8 to 89.9] | 88.8 [85.1 to 92.5]
  Week 20 | 88.4 [84.6 to 92.2] | 90.3 [86.8 to 93.7]
  Week 24 | 90.9 [87.6 to 94.3] | 89.6 [86.0 to 93.1]

7. Secondary Outcome: Part 1: Percentage of Participants Gaining >0 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 90.2 [86.8 to 93.6] | 93.2 [90.3 to 96.1]
  Week 8 | 92.7 [89.7 to 95.8] | 96.8 [94.7 to 98.8]
  Week 12 | 94.9 [92.4 to 97.5] | 94.2 [91.5 to 97.0]
  Week 16 | 93.8 [91.1 to 96.6] | 94.9 [92.4 to 97.5]
  Week 20 | 94.9 [92.4 to 97.5] | 96.0 [93.8 to 98.3]
  Week 24 | 96.4 [94.2 to 98.6] | 95.3 [92.9 to 97.8]

8. Secondary Outcome: Part 1: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 99.3 [98.3 to 100.0] | 98.9 [97.7 to 100.0]
  Week 8 | 99.3 [98.3 to 100.0] | 98.9 [97.7 to 100.0]
  Week 12 | 99.3 [98.3 to 100.0] | 98.9 [97.7 to 100.0]
  Week 16 | 99.3 [98.3 to 100.0] | 98.6 [97.2 to 99.9]
  Week 20 | 99.6 [98.9 to 100.0] | 98.6 [97.2 to 99.9]
  Week 24 | 99.6 [98.9 to 100.0] | 98.6 [97.2 to 99.9]

9. Secondary Outcome: Part 1: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 98.5 [97.1 to 99.9] | 98.9 [97.7 to 100.0]
  Week 8 | 98.5 [97.1 to 100.0] | 98.9 [97.7 to 100.0]
  Week 12 | 98.5 [97.1 to 99.9] | 98.9 [97.7 to 100.0]
  Week 16 | 98.5 [97.1 to 99.9] | 98.2 [96.7 to 99.7]
  Week 20 | 99.3 [98.3 to 100.0] | 98.6 [97.2 to 99.9]
  Week 24 | 99.6 [98.9 to 100.0] | 98.2 [96.7 to 99.7]

10. Secondary Outcome: Part 1: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 97.1 [95.1 to 99.1] | 98.6 [97.2 to 99.9]
  Week 8 | 97.8 [96.1 to 99.5] | 98.6 [97.2 to 99.9]
  Week 12 | 97.8 [96.1 to 99.5] | 98.9 [97.7 to 100.0]
  Week 16 | 97.8 [96.1 to 99.5] | 98.2 [96.7 to 99.7]
  Week 20 | 98.5 [97.1 to 99.9] | 97.8 [96.2 to 99.5]
  Week 24 | 98.6 [97.2 to 100.0] | 97.5 [95.7 to 99.3]

11. Secondary Outcome: Part 1: Percentage of Participants Achieving ≥84 Letters in BCVA (20/20 Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 8.7 [5.5 to 11.9] | 8.6 [5.5 to 11.8]
  Week 8 | 14.1 [10.3 to 18.0] | 15.5 [11.5 to 19.5]
  Week 12 | 15.6 [11.7 to 19.6] | 20.2 [15.7 to 24.6]
  Week 16 | 17.4 [13.3 to 21.6] | 22.0 [17.4 to 26.5]
  Week 20 | 20.7 [16.2 to 25.2] | 23.8 [19.0 to 28.5]
  Week 24 | 22.9 [18.2 to 27.6] | 23.8 [19.1 to 28.5]

12. Secondary Outcome: Part 1: Percentage of Participants Achieving ≥69 Letters in BCVA (20/40 or Better Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 55.6 [50.6 to 60.5] | 62.3 [57.3 to 67.3]
  Week 8 | 63.9 [59.3 to 68.6] | 70.3 [65.7 to 74.9]
  Week 12 | 69.0 [64.4 to 73.6] | 69.2 [64.4 to 74.0]
  Week 16 | 72.2 [67.7 to 76.8] | 72.1 [67.5 to 76.8]
  Week 20 | 73.3 [69.1 to 77.6] | 76.1 [71.7 to 80.5]
  Week 24 | 73.7 [69.3 to 78.1] | 76.5 [71.9 to 81.0]

13. Secondary Outcome: Part 1: Percentage of Participants With ≤38 Letters in BCVA (20/200 or Worse Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 24
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (>38 and ≤38 letters) and region (U.S. and Canada, Asia, and rest of the world). All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 3.6 [2.0 to 5.3] | 1.5 [0.1 to 2.9]
  Week 8 | 3.2 [1.3 to 5.0] | 1.9 [0.5 to 3.3]
  Week 12 | 2.3 [0.8 to 3.8] | 1.5 [0.2 to 2.8]
  Week 16 | 2.3 [0.8 to 3.8] | 1.9 [0.4 to 3.3]
  Week 20 | 2.3 [0.8 to 3.8] | 1.9 [0.4 to 3.3]
  Week 24 | 2.3 [0.8 to 3.8] | 1.9 [0.4 to 3.3]

14. Secondary Outcome: Part 1: Change From Baseline in Central Subfield Thickness in the Study Eye at Specified Timepoints Through Week 24
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) using optical coherence tomography (OCT), as assessed by the central reading center. The Mixed Model of Repeated Measures (MMRM) analysis included the categorical covariates of treatment arm, visit, visit-by-treatment arm interaction, baseline CST (continuous), and randomization stratification factors [baseline BCVA (≥55 and ≤54 letters), and region (U.S. and Canada, Asia, and rest of the world)] as fixed effects. An unstructured covariance structure was used. Missing data were implicitly imputed by MMRM model assuming missing at random. Treatment policy strategy (i.e., all observed values used) was applied to all intercurrent events (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
microns
  Week 4 | -283.9 [-290.1 to -277.8] | -281.1 [-287.2 to -274.9]
  Week 8 | -299.4 [-305.2 to -293.7] | -296.9 [-302.6 to -291.2]
  Week 12 | -304.4 [-309.7 to -299.1] | -298.8 [-304.1 to -293.5]
  Week 16 | -306.1 [-311.5 to -300.8] | -301.4 [-306.7 to -296.1]
  Week 20 | -307.3 [-312.5 to -302.1] | -302.2 [-307.4 to -297.0]
  Week 24 | -311.4 [-316.4 to -306.4] | -304.4 [-309.3 to -299.4]

15. Secondary Outcome: Part 1: Percentage of Participants With Absence of Macular Edema in the Study Eye at Specified Timepoints Through Week 24
Description: Absence of diabetic macular edema was defined as achieving a central subfield thickness of <325 microns in the study eye. Central subfield thickness was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≥55 and ≤54 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 88.8 [85.1 to 92.5] | 88.1 [84.4 to 91.9]
  Week 8 | 94.5 [91.9 to 97.2] | 93.2 [90.3 to 96.1]
  Week 12 | 96.4 [94.2 to 98.5] | 92.1 [89.0 to 95.2]
  Week 16 | 95.3 [92.8 to 97.7] | 93.6 [90.7 to 96.4]
  Week 20 | 96.0 [93.7 to 98.3] | 94.6 [92.1 to 97.2]
  Week 24 | 95.3 [92.8 to 97.7] | 93.9 [91.2 to 96.6]

16. Secondary Outcome: Part 1: Percentage of Participants With Absence of Intraretinal Fluid in the Study Eye at Specified Timepoints Through Week 24
Description: Intraretinal fluid was measured in the study eye using optical coherence tomography (OCT) in the central subfield (center 1 mm) by a central reading center. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≥55 and ≤54 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 46.1 [40.2 to 51.9] | 54.8 [49.0 to 60.6]
  Week 8 | 53.8 [48.2 to 59.4] | 57.4 [51.6 to 63.1]
  Week 12 | 65.3 [59.7 to 70.8] | 56.6 [50.8 to 62.4]
  Week 16 | 69.9 [64.6 to 75.3] | 72.9 [67.8 to 78.1]
  Week 20 | 67.1 [61.6 to 72.6] | 66.4 [60.9 to 71.9]
  Week 24 | 72.5 [67.3 to 77.7] | 66.0 [60.5 to 71.6]

17. Secondary Outcome: Part 1: Percentage of Participants With Absence of Subretinal Fluid in the Study Eye at Specified Timepoints Through Week 24
Description: Subretinal fluid was measured in the study eye using optical coherence tomography (OCT) in the central subfield (center 1 mm) by a central reading center. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≥55 and ≤54 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 76.1 [71.1 to 81.1] | 72.9 [67.8 to 78.1]
  Week 8 | 93.1 [90.2 to 96.1] | 91.4 [88.1 to 94.6]
  Week 12 | 96.4 [94.2 to 98.6] | 97.1 [95.2 to 99.1]
  Week 16 | 95.3 [92.8 to 97.8] | 96.4 [94.2 to 98.6]
  Week 20 | 98.2 [96.6 to 99.8] | 97.8 [96.1 to 99.5]
  Week 24 | 91.3 [88.0 to 94.6] | 90.3 [86.9 to 93.7]

18. Secondary Outcome: Part 1: Percentage of Participants With Absence of Intraretinal Fluid and Subretinal Fluid in the Study Eye at Specified Timepoints Through Week 24
Description: Intraretinal fluid and subretinal fluid were measured in the study eye using optical coherence tomography (OCT) in the central subfield (center 1 mm) by a central reading center. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≥55 and ≤54 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 37.8 [32.1 to 43.4] | 40.8 [35.2 to 46.4]
  Week 8 | 50.9 [45.3 to 56.5] | 54.1 [48.4 to 59.9]
  Week 12 | 63.8 [58.2 to 69.4] | 56.3 [50.5 to 62.1]
  Week 16 | 67.1 [61.6 to 72.6] | 72.6 [67.4 to 77.8]
  Week 20 | 66.0 [60.5 to 71.5] | 66.0 [60.5 to 71.6]
  Week 24 | 66.3 [60.8 to 71.9] | 61.0 [55.3 to 66.7]

19. Secondary Outcome: Part 1: Change From Baseline in National Eye Institute 25-Item Visual Functioning Questionnaire (NEI VFQ-25) Composite Score at Week 24
Description: The NEI VFQ-25 captures a patient's perception of vision-related functioning and vision-related quality of life. The core measure includes 25 items that comprise 11 vision-related subscales and 1 item on general health. The composite score ranges from 0 to 100, with higher scores indicating better vision-related functioning. For the ANCOVA analysis, the model uses the non-missing change from baseline in BCVA at Weeks 24 as the response variables adjusted for the treatment group, baseline NEI VFQ-25 Composite Score (continuous), baseline BCVA score (≥55 and ≤54 letters) and region (U.S. and Canada, Asia, and the rest of the world). Observed NEI VFQ-25 assessments were used regardless of the occurrence of intercurrent events. Missing data were not imputed. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with non-missing Baseline and Week 24 assessments were included for analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 253 | 244
score on a scale | 5.6 [4.5 to 6.7] | 5.9 [4.8 to 7.1]
Statistical Analysis 1: Comparison: Arm A: Faricimab Q4W (Part 1) vs Arm B: Aflibercept Q4W (Part 1); Test type: Other; Difference in Adjusted Means = -0.4, 95% CI 2-sided [-1.9 to 1.1], Standard Error of Mean 0.76

20. Secondary Outcome: Parts 1 and 2: Change From Baseline in BCVA in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
ETDRS Letters
  Week 4 | 11.5 [10.5 to 12.5] | 12.4 [11.4 to 13.4]
  Week 8 | 13.7 [12.6 to 14.7] | 15.1 [14.1 to 16.2]
  Week 12 | 15.1 [14.0 to 16.1] | 15.9 [14.8 to 17.0]
  Week 16 | 15.5 [14.4 to 16.6] | 16.5 [15.4 to 17.6]
  Week 20 | 16.3 [15.1 to 17.4] | 17.2 [16.1 to 18.4]
  Week 24 | 16.8 [15.6 to 17.9] | 17.5 [16.3 to 18.6]
  Week 28 | 16.5 [15.3 to 17.6] | 17.3 [16.2 to 18.4]
  Week 32 | 17.2 [16.0 to 18.4] | 17.5 [16.3 to 18.7]
  Week 36 | 17.3 [16.1 to 18.4] | 18.0 [16.8 to 19.2]
  Week 40 | 17.3 [16.1 to 18.4] | 17.7 [16.6 to 18.9]
  Week 44 | 18.1 [16.8 to 19.3] | 17.7 [16.5 to 18.9]
  Week 48 | 18.0 [16.8 to 19.3] | 18.2 [17.0 to 19.4]
  Week 52 | 18.0 [16.7 to 19.3] | 18.4 [17.1 to 19.7]
  Week 56 | 17.3 [16.0 to 18.6] | 18.1 [16.8 to 19.4]
  Week 60 | 18.0 [16.7 to 19.3] | 18.6 [17.3 to 19.8]
  Week 64 | 17.9 [16.6 to 19.2] | 18.6 [17.3 to 19.9]
  Week 68 | 18.1 [16.8 to 19.4] | 18.8 [17.5 to 20.1]
  Week 72 | 18.4 [17.1 to 19.7] | 18.8 [17.5 to 20.1]

21. Secondary Outcome: Parts 1 and 2: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 34.3 [28.9 to 39.8] | 36.9 [31.5 to 42.3]
  Week 8 | 41.2 [35.6 to 46.9] | 46.7 [41.0 to 52.3]
  Week 12 | 51.0 [45.3 to 56.7] | 52.1 [46.3 to 57.8]
  Week 16 | 53.6 [47.8 to 59.3] | 56.4 [50.8 to 62.1]
  Week 20 | 56.1 [50.3 to 61.8] | 58.9 [53.3 to 64.6]
  Week 24 | 56.1 [50.4 to 61.9] | 60.4 [54.7 to 66.0]
  Week 28 | 55.8 [50.0 to 61.5] | 61.8 [56.2 to 67.4]
  Week 32 | 59.0 [53.3 to 64.6] | 61.4 [55.8 to 67.1]
  Week 36 | 61.2 [55.5 to 66.8] | 62.5 [56.9 to 68.1]
  Week 40 | 60.8 [55.2 to 66.4] | 61.1 [55.4 to 66.7]
  Week 44 | 65.5 [60.1 to 71.0] | 58.9 [53.4 to 64.5]
  Week 48 | 64.1 [58.5 to 69.6] | 60.7 [55.1 to 66.3]
  Week 52 | 61.2 [55.6 to 66.8] | 64.0 [58.4 to 69.5]
  Week 56 | 57.9 [52.3 to 63.5] | 63.6 [58.1 to 69.2]
  Week 60 | 62.6 [57.1 to 68.1] | 62.9 [57.4 to 68.4]
  Week 64 | 61.9 [56.3 to 67.4] | 65.4 [59.9 to 70.9]
  Week 68 | 63.0 [57.5 to 68.4] | 64.7 [59.2 to 70.2]
  Week 72 | 62.3 [56.7 to 67.8] | 66.9 [61.5 to 72.3]

22. Secondary Outcome: Parts 1 and 2: Percentage of Participants Gaining ≥10 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 57.5 [51.8 to 63.3] | 59.2 [53.6 to 64.9]
  Week 8 | 69.1 [63.8 to 74.5] | 69.0 [63.6 to 74.4]
  Week 12 | 75.0 [69.9 to 80.1] | 74.8 [69.7 to 79.8]
  Week 16 | 72.1 [66.9 to 77.3] | 76.6 [71.6 to 81.5]
  Week 20 | 75.3 [70.3 to 80.4] | 79.1 [74.3 to 83.9]
  Week 24 | 77.5 [72.6 to 82.4] | 77.3 [72.4 to 82.2]
  Week 28 | 76.1 [71.1 to 81.1] | 76.6 [71.6 to 81.5]
  Week 32 | 77.5 [72.6 to 82.4] | 78.4 [73.6 to 83.2]
  Week 36 | 75.7 [70.7 to 80.7] | 78.7 [74.0 to 83.5]
  Week 40 | 77.5 [72.7 to 82.4] | 76.2 [71.3 to 81.2]
  Week 44 | 80.4 [75.8 to 85.1] | 76.6 [71.7 to 81.5]
  Week 48 | 79.7 [75.0 to 84.4] | 79.4 [74.7 to 84.2]
  Week 52 | 80.8 [76.2 to 85.4] | 80.2 [75.5 to 84.8]
  Week 56 | 75.7 [70.7 to 80.7] | 78.0 [73.2 to 82.9]
  Week 60 | 79.3 [74.6 to 84.0] | 80.5 [75.9 to 85.2]
  Week 64 | 78.9 [74.2 to 83.7] | 78.7 [73.9 to 83.5]
  Week 68 | 78.9 [74.2 to 83.7] | 77.3 [72.4 to 82.2]
  Week 72 | 80.4 [75.8 to 85.0] | 79.5 [74.7 to 84.2]

23. Secondary Outcome: Parts 1 and 2: Percentage of Participants Gaining ≥5 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 75.7 [70.7 to 80.7] | 79.1 [74.4 to 83.9]
  Week 8 | 84.0 [79.7 to 88.3] | 88.1 [84.3 to 91.9]
  Week 12 | 87.0 [83.1 to 90.9] | 87.0 [83.1 to 91.0]
  Week 16 | 85.9 [81.8 to 89.9] | 88.8 [85.1 to 92.5]
  Week 20 | 88.4 [84.6 to 92.2] | 90.3 [86.8 to 93.7]
  Week 24 | 90.9 [87.6 to 94.3] | 89.6 [86.0 to 93.1]
  Week 28 | 89.1 [85.5 to 92.8] | 87.8 [84.0 to 91.6]
  Week 32 | 89.5 [85.9 to 93.1] | 87.7 [83.9 to 91.6]
  Week 36 | 88.4 [84.6 to 92.1] | 90.6 [87.2 to 94.0]
  Week 40 | 90.2 [86.7 to 93.7] | 90.6 [87.2 to 94.0]
  Week 44 | 89.1 [85.5 to 92.8] | 88.4 [84.7 to 92.2]
  Week 48 | 88.4 [84.6 to 92.2] | 90.3 [86.8 to 93.8]
  Week 52 | 89.9 [86.4 to 93.4] | 88.5 [84.7 to 92.2]
  Week 56 | 88.0 [84.3 to 91.8] | 87.0 [83.1 to 91.0]
  Week 60 | 89.9 [86.3 to 93.4] | 88.1 [84.3 to 91.9]
  Week 64 | 90.6 [87.1 to 94.0] | 87.7 [83.9 to 91.6]
  Week 68 | 89.5 [85.9 to 93.1] | 87.1 [83.1 to 91.0]
  Week 72 | 89.8 [86.3 to 93.4] | 87.4 [83.5 to 91.3]

24. Secondary Outcome: Parts 1 and 2: Percentage of Participants Gaining >0 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 90.2 [86.8 to 93.6] | 93.2 [90.3 to 96.1]
  Week 8 | 92.7 [89.7 to 95.8] | 96.8 [94.7 to 98.8]
  Week 12 | 94.9 [92.4 to 97.5] | 94.2 [91.5 to 97.0]
  Week 16 | 93.8 [91.1 to 96.6] | 94.9 [92.4 to 97.5]
  Week 20 | 94.9 [92.4 to 97.5] | 96.0 [93.8 to 98.3]
  Week 24 | 96.4 [94.2 to 98.6] | 95.3 [92.9 to 97.8]
  Week 28 | 95.3 [92.9 to 97.8] | 95.0 [92.4 to 97.5]
  Week 32 | 96.0 [93.8 to 98.3] | 95.0 [92.4 to 97.5]
  Week 36 | 94.2 [91.5 to 96.9] | 94.6 [92.0 to 97.2]
  Week 40 | 94.6 [91.9 to 97.2] | 95.7 [93.3 to 98.0]
  Week 44 | 95.3 [92.9 to 97.7] | 94.6 [92.0 to 97.2]
  Week 48 | 94.6 [92.0 to 97.2] | 96.1 [93.8 to 98.3]
  Week 52 | 93.8 [91.1 to 96.6] | 94.6 [92.1 to 97.2]
  Week 56 | 93.1 [90.2 to 96.1] | 95.3 [92.9 to 97.8]
  Week 60 | 94.6 [91.9 to 97.2] | 94.2 [91.5 to 97.0]
  Week 64 | 94.9 [92.4 to 97.5] | 94.2 [91.5 to 97.0]
  Week 68 | 93.5 [90.6 to 96.4] | 93.9 [91.1 to 96.7]
  Week 72 | 94.6 [91.9 to 97.2] | 93.9 [91.1 to 96.7]

25. Secondary Outcome: Parts 1 and 2: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 99.3 [98.3 to 100.0] | 98.9 [97.7 to 100.0]
  Week 8 | 99.3 [98.3 to 100.0] | 98.9 [97.7 to 100.0]
  Week 12 | 99.3 [98.3 to 100.0] | 98.9 [97.7 to 100.0]
  Week 16 | 99.3 [98.3 to 100.0] | 98.6 [97.2 to 99.9]
  Week 20 | 99.6 [98.9 to 100.0] | 98.6 [97.2 to 99.9]
  Week 24 | 99.6 [98.9 to 100.0] | 98.6 [97.2 to 99.9]
  Week 28 | 99.6 [98.9 to 100.0] | 98.6 [97.2 to 99.9]
  Week 32 | 99.6 [98.9 to 100.0] | 98.6 [97.2 to 99.9]
  Week 36 | 99.6 [98.9 to 100.0] | 98.6 [97.2 to 100.0]
  Week 40 | 98.9 [97.7 to 100.0] | 98.6 [97.2 to 100.0]
  Week 44 | 99.3 [98.3 to 100.0] | 98.6 [97.2 to 100.0]
  Week 48 | 99.3 [98.3 to 100.0] | 98.2 [96.7 to 99.8]
  Week 52 | 98.6 [97.2 to 100.0] | 98.2 [96.7 to 99.8]
  Week 56 | 98.9 [97.7 to 100.0] | 98.2 [96.7 to 99.8]
  Week 60 | 99.3 [98.3 to 100.0] | 98.2 [96.7 to 99.8]
  Week 64 | 98.9 [97.7 to 100.0] | 97.9 [96.2 to 99.5]
  Week 68 | 98.9 [97.7 to 100.0] | 98.2 [96.7 to 99.8]
  Week 72 | 98.9 [97.7 to 100.0] | 98.2 [96.7 to 99.8]

26. Secondary Outcome: Parts 1 and 2: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 98.5 [97.1 to 99.9] | 98.9 [97.7 to 100.0]
  Week 8 | 98.5 [97.1 to 100.0] | 98.9 [97.7 to 100.0]
  Week 12 | 98.5 [97.1 to 99.9] | 98.9 [97.7 to 100.0]
  Week 16 | 98.5 [97.1 to 99.9] | 98.2 [96.7 to 99.7]
  Week 20 | 99.3 [98.3 to 100.0] | 98.6 [97.2 to 99.9]
  Week 24 | 99.6 [98.9 to 100.0] | 98.2 [96.7 to 99.7]
  Week 28 | 99.6 [98.9 to 100.0] | 98.2 [96.7 to 99.7]
  Week 32 | 99.3 [98.3 to 100.0] | 98.2 [96.7 to 99.7]
  Week 36 | 99.6 [98.9 to 100.0] | 98.6 [97.2 to 100.0]
  Week 40 | 98.9 [97.7 to 100.0] | 98.6 [97.2 to 100.0]
  Week 44 | 99.3 [98.3 to 100.0] | 98.2 [96.7 to 99.8]
  Week 48 | 98.9 [97.7 to 100.0] | 98.2 [96.7 to 99.8]
  Week 52 | 98.6 [97.2 to 100.0] | 98.2 [96.7 to 99.8]
  Week 56 | 98.9 [97.7 to 100.0] | 97.9 [96.2 to 99.5]
  Week 60 | 98.9 [97.7 to 100.0] | 98.2 [96.7 to 99.8]
  Week 64 | 98.6 [97.2 to 99.9] | 97.1 [95.2 to 99.1]
  Week 68 | 98.6 [97.2 to 100.0] | 97.9 [96.2 to 99.5]
  Week 72 | 98.2 [96.6 to 99.8] | 97.9 [96.2 to 99.5]

27. Secondary Outcome: Parts 1 and 2: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 97.1 [95.1 to 99.1] | 98.6 [97.2 to 99.9]
  Week 8 | 97.8 [96.1 to 99.5] | 98.6 [97.2 to 99.9]
  Week 12 | 97.8 [96.1 to 99.5] | 98.9 [97.7 to 100.0]
  Week 16 | 97.8 [96.1 to 99.5] | 98.2 [96.7 to 99.7]
  Week 20 | 98.5 [97.1 to 99.9] | 97.8 [96.2 to 99.5]
  Week 24 | 98.6 [97.2 to 100.0] | 97.5 [95.7 to 99.3]
  Week 28 | 98.2 [96.6 to 99.8] | 97.5 [95.7 to 99.3]
  Week 32 | 98.6 [97.2 to 99.9] | 97.8 [96.2 to 99.5]
  Week 36 | 98.2 [96.7 to 99.7] | 97.5 [95.7 to 99.3]
  Week 40 | 97.1 [95.2 to 99.0] | 97.5 [95.6 to 99.3]
  Week 44 | 98.6 [97.2 to 99.9] | 97.8 [96.1 to 99.5]
  Week 48 | 97.1 [95.2 to 99.0] | 97.9 [96.2 to 99.5]
  Week 52 | 97.1 [95.2 to 99.1] | 97.5 [95.7 to 99.3]
  Week 56 | 97.5 [95.6 to 99.3] | 97.5 [95.7 to 99.3]
  Week 60 | 97.8 [96.1 to 99.5] | 96.8 [94.7 to 98.8]
  Week 64 | 97.1 [95.1 to 99.1] | 96.8 [94.7 to 98.8]
  Week 68 | 97.1 [95.1 to 99.1] | 97.1 [95.2 to 99.1]
  Week 72 | 97.1 [95.1 to 99.1] | 96.8 [94.7 to 98.8]

28. Secondary Outcome: Parts 1 and 2: Percentage of Participants Achieving ≥84 Letters in BCVA (20/20 Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 8.7 [5.5 to 11.9] | 8.6 [5.5 to 11.8]
  Week 8 | 14.1 [10.3 to 18.0] | 15.5 [11.5 to 19.5]
  Week 12 | 15.6 [11.7 to 19.6] | 20.2 [15.7 to 24.6]
  Week 16 | 17.4 [13.3 to 21.6] | 22.0 [17.4 to 26.5]
  Week 20 | 20.7 [16.2 to 25.2] | 23.8 [19.0 to 28.5]
  Week 24 | 22.9 [18.2 to 27.6] | 23.8 [19.1 to 28.5]
  Week 28 | 24.0 [19.2 to 28.8] | 25.6 [20.7 to 30.4]
  Week 32 | 25.1 [20.3 to 29.8] | 23.4 [18.8 to 28.0]
  Week 36 | 25.1 [20.2 to 29.9] | 25.2 [20.4 to 30.0]
  Week 40 | 26.9 [22.0 to 31.8] | 22.0 [17.4 to 26.5]
  Week 44 | 26.8 [21.8 to 31.8] | 24.8 [20.0 to 29.7]
  Week 48 | 29.0 [24.0 to 34.1] | 25.2 [20.3 to 30.1]
  Week 52 | 26.8 [21.9 to 31.7] | 25.6 [20.7 to 30.4]
  Week 56 | 26.1 [21.2 to 31.0] | 22.0 [17.3 to 26.6]
  Week 60 | 27.6 [22.6 to 32.6] | 25.6 [20.8 to 30.4]
  Week 64 | 30.1 [25.0 to 35.3] | 24.5 [19.7 to 29.3]
  Week 68 | 29.4 [24.2 to 34.6] | 25.9 [21.0 to 30.8]
  Week 72 | 29.4 [24.3 to 34.5] | 24.8 [20.0 to 29.7]

29. Secondary Outcome: Parts 1 and 2: Percentage of Participants Achieving ≥69 Letters in BCVA (20/40 or Better Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 55.6 [50.6 to 60.5] | 62.3 [57.3 to 67.3]
  Week 8 | 63.9 [59.3 to 68.6] | 70.3 [65.7 to 74.9]
  Week 12 | 69.0 [64.4 to 73.6] | 69.2 [64.4 to 74.0]
  Week 16 | 72.2 [67.7 to 76.8] | 72.1 [67.5 to 76.8]
  Week 20 | 73.3 [69.1 to 77.6] | 76.1 [71.7 to 80.5]
  Week 24 | 73.7 [69.3 to 78.1] | 76.5 [71.9 to 81.0]
  Week 28 | 73.3 [68.7 to 77.9] | 75.4 [70.7 to 80.0]
  Week 32 | 76.9 [72.6 to 81.2] | 75.4 [70.7 to 80.1]
  Week 36 | 76.2 [71.8 to 80.6] | 77.9 [73.3 to 82.5]
  Week 40 | 75.5 [71.0 to 79.9] | 76.8 [72.3 to 81.3]
  Week 44 | 76.9 [72.4 to 81.4] | 76.1 [71.4 to 80.7]
  Week 48 | 77.2 [72.7 to 81.8] | 79.3 [75.0 to 83.7]
  Week 52 | 78.7 [74.3 to 83.1] | 80.4 [76.1 to 84.7]
  Week 56 | 76.2 [71.5 to 80.9] | 79.0 [74.5 to 83.5]
  Week 60 | 80.2 [75.8 to 84.5] | 79.0 [74.5 to 83.5]
  Week 64 | 77.6 [73.0 to 82.2] | 81.1 [76.8 to 85.5]
  Week 68 | 77.6 [73.0 to 82.2] | 80.4 [76.0 to 84.9]
  Week 72 | 78.0 [73.5 to 82.4] | 79.0 [74.4 to 83.6]

30. Secondary Outcome: Parts 1 and 2: Percentage of Participants With ≤38 Letters in BCVA (20/200 or Worse Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 13
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 3.6 [2.0 to 5.3] | 1.5 [0.1 to 2.9]
  Week 8 | 3.2 [1.3 to 5.0] | 1.9 [0.5 to 3.3]
  Week 12 | 2.3 [0.8 to 3.8] | 1.5 [0.2 to 2.8]
  Week 16 | 2.3 [0.8 to 3.8] | 1.9 [0.4 to 3.3]
  Week 20 | 2.3 [0.8 to 3.8] | 1.9 [0.4 to 3.3]
  Week 24 | 2.3 [0.8 to 3.8] | 1.9 [0.4 to 3.3]
  Week 28 | 2.0 [0.6 to 3.5] | 1.9 [0.4 to 3.3]
  Week 32 | 2.4 [0.8 to 4.0] | 1.9 [0.4 to 3.3]
  Week 36 | 1.9 [0.5 to 3.4] | 1.5 [0.2 to 2.8]
  Week 40 | 2.3 [0.8 to 3.7] | 1.5 [0.2 to 2.8]
  Week 44 | 2.7 [1.0 to 4.4] | 1.5 [0.2 to 2.8]
  Week 48 | 2.4 [0.8 to 4.0] | 2.2 [0.6 to 3.9]
  Week 52 | 3.1 [1.3 to 4.9] | 2.6 [0.9 to 4.3]
  Week 56 | 2.7 [1.0 to 4.4] | 2.6 [0.9 to 4.3]
  Week 60 | 2.1 [0.6 to 3.6] | 2.6 [0.9 to 4.3]
  Week 64 | 3.1 [1.3 to 4.9] | 2.2 [0.6 to 3.9]
  Week 68 | 2.1 [0.6 to 3.6] | 1.8 [0.3 to 3.3]
  Week 72 | 2.1 [0.6 to 3.6] | 2.2 [0.5 to 3.9]

31. Secondary Outcome: Parts 1 and 2: Change From Baseline in NEI VFQ-25 Questionnaire Composite Score at Specified Timepoints Through Week 72
Description: The NEI VFQ-25 captures a patient's perception of vision-related functioning and vision-related quality of life. The core measure includes 25 items that comprise 11 vision-related subscales and 1 item on general health. The composite score ranges from 0 to 100, with higher scores indicating better vision-related functioning. For the MMRM analysis, the model adjusted for the treatment group, visit, visit-by-treatment group interaction, baseline NEI VFQ-25 Composite Score continuous), baseline BCVA score (≥55 and ≤54 letters), and region (U.S. and Canada, Asia, and the rest of the world). Observed NEI VFQ-25 assessments were used regardless of the occurrence of intercurrent events. Missing data were implicitly imputed. Invalid BCVA values were excluded. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline and Weeks 24, 48, and 72
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
score on a scale
  Week 24 | 5.6 [4.5 to 6.6] | 5.9 [4.9 to 7.0]
  Week 48 | 6.4 [5.3 to 7.5] | 6.3 [5.2 to 7.4]
  Week 72 | 6.0 [4.8 to 7.3] | 7.8 [6.6 to 9.0]

32. Secondary Outcome: Parts 1 and 2: Change From Baseline in Central Subfield Thickness in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 14
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
microns
  Week 4 | -287.3 [-293.5 to -281.1] | -284.3 [-290.4 to -278.2]
  Week 8 | -302.9 [-308.7 to -297.2] | -300.2 [-306.0 to -294.5]
  Week 12 | -307.8 [-313.1 to -302.6] | -301.9 [-307.1 to -296.7]
  Week 16 | -309.3 [-314.6 to -304.0] | -304.5 [-309.8 to -299.3]
  Week 20 | -310.6 [-315.5 to -305.6] | -304.2 [-309.1 to -299.3]
  Week 24 | -314.5 [-319.5 to -309.6] | -307.6 [-312.5 to -302.7]
  Week 28 | -294.0 [-302.2 to -285.8] | -285.1 [-293.3 to -276.9]
  Week 32 | -308.3 [-314.6 to -302.0] | -303.2 [-309.4 to -297.0]
  Week 36 | -304.1 [-310.6 to -297.6] | -298.8 [-305.2 to -292.4]
  Week 40 | -296.7 [-304.4 to -288.9] | -285.8 [-293.7 to -278.0]
  Week 44 | -309.2 [-315.9 to -302.5] | -301.6 [-308.3 to -294.9]
  Week 48 | -309.4 [-315.3 to -303.5] | -302.8 [-308.7 to -296.9]
  Week 52 | -302.2 [-308.6 to -295.7] | -302.4 [-308.8 to -296.0]
  Week 56 | -294.0 [-302.6 to -285.5] | -288.0 [-296.6 to -279.4]
  Week 60 | -309.5 [-315.1 to -303.9] | -306.2 [-311.9 to -300.6]
  Week 64 | -311.1 [-316.3 to -305.9] | -305.9 [-311.1 to -300.7]
  Week 68 | -311.2 [-316.3 to -306.1] | -307.9 [-313.0 to -302.8]
  Week 72 | -310.5 [-315.7 to -305.4] | -307.2 [-312.3 to -302.0]

33. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Absence of Macular Edema in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 15
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 88.8 [85.1 to 92.5] | 88.1 [84.4 to 91.9]
  Week 8 | 94.5 [91.9 to 97.2] | 93.2 [90.3 to 96.1]
  Week 12 | 96.4 [94.2 to 98.5] | 92.1 [89.0 to 95.2]
  Week 16 | 95.3 [92.8 to 97.7] | 93.6 [90.7 to 96.4]
  Week 20 | 96.0 [93.7 to 98.3] | 94.6 [92.1 to 97.2]
  Week 24 | 95.6 [93.3 to 98.0] | 94.3 [91.6 to 96.9]
  Week 28 | 89.1 [85.5 to 92.8] | 86.0 [82.0 to 90.0]
  Week 32 | 94.6 [91.9 to 97.2] | 92.5 [89.4 to 95.5]
  Week 36 | 93.8 [91.1 to 96.5] | 90.7 [87.3 to 94.0]
  Week 40 | 89.5 [85.9 to 93.0] | 84.2 [79.9 to 88.4]
  Week 44 | 96.0 [93.7 to 98.3] | 92.1 [88.9 to 95.2]
  Week 48 | 94.9 [92.4 to 97.5] | 91.4 [88.1 to 94.6]
  Week 52 | 92.4 [89.3 to 95.5] | 91.4 [88.2 to 94.6]
  Week 56 | 89.5 [85.9 to 93.1] | 86.3 [82.3 to 90.3]
  Week 60 | 94.2 [91.5 to 96.9] | 93.9 [91.1 to 96.7]
  Week 64 | 95.3 [92.8 to 97.8] | 93.9 [91.1 to 96.7]
  Week 68 | 94.9 [92.4 to 97.5] | 92.4 [89.4 to 95.5]
  Week 72 | 94.2 [91.5 to 96.9] | 94.2 [91.5 to 97.0]

34. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Absence of Intraretinal Fluid in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 16
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 46.1 [40.2 to 51.9] | 54.8 [49.0 to 60.6]
  Week 8 | 53.8 [48.2 to 59.4] | 57.4 [51.6 to 63.1]
  Week 12 | 65.3 [59.7 to 70.8] | 56.6 [50.8 to 62.4]
  Week 16 | 69.9 [64.6 to 75.3] | 72.9 [67.8 to 78.1]
  Week 20 | 67.1 [61.6 to 72.6] | 66.4 [60.9 to 71.9]
  Week 24 | 73.9 [68.9 to 79.0] | 69.3 [63.9 to 74.7]
  Week 28 | 54.4 [48.7 to 60.2] | 47.6 [41.8 to 53.5]
  Week 32 | 68.1 [62.6 to 73.6] | 65.0 [59.4 to 70.6]
  Week 36 | 60.9 [55.1 to 66.6] | 56.0 [50.2 to 61.7]
  Week 40 | 50.8 [45.0 to 56.6] | 48.1 [42.3 to 53.9]
  Week 44 | 70.3 [64.9 to 75.6] | 63.9 [58.3 to 69.6]
  Week 48 | 76.1 [71.1 to 81.1] | 67.9 [62.5 to 73.3]
  Week 52 | 55.8 [50.0 to 61.7] | 56.7 [50.9 to 62.5]
  Week 56 | 58.4 [52.6 to 64.1] | 58.9 [53.2 to 64.6]
  Week 60 | 75.0 [69.9 to 80.1] | 72.6 [67.4 to 77.7]
  Week 64 | 75.8 [70.9 to 80.7] | 69.7 [64.3 to 75.1]
  Week 68 | 69.9 [64.5 to 75.3] | 68.6 [63.2 to 74.1]
  Week 72 | 72.8 [67.6 to 78.0] | 72.9 [67.7 to 78.1]

35. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Absence of Subretinal Fluid in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 17
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 76.1 [71.1 to 81.1] | 72.9 [67.8 to 78.1]
  Week 8 | 93.1 [90.2 to 96.1] | 91.4 [88.1 to 94.6]
  Week 12 | 96.4 [94.2 to 98.6] | 97.1 [95.2 to 99.1]
  Week 16 | 95.3 [92.8 to 97.8] | 96.4 [94.2 to 98.6]
  Week 20 | 98.2 [96.6 to 99.8] | 97.8 [96.1 to 99.5]
  Week 24 | 91.3 [88.0 to 94.6] | 90.3 [86.9 to 93.7]
  Week 28 | 93.5 [90.7 to 96.4] | 91.0 [87.6 to 94.3]
  Week 32 | 96.4 [94.2 to 98.6] | 97.1 [95.2 to 99.1]
  Week 36 | 97.1 [95.1 to 99.1] | 96.0 [93.7 to 98.3]
  Week 40 | 96.8 [94.7 to 98.8] | 95.7 [93.3 to 98.1]
  Week 44 | 97.5 [95.7 to 99.3] | 95.7 [93.3 to 98.0]
  Week 48 | 97.1 [95.1 to 99.1] | 94.6 [91.9 to 97.2]
  Week 52 | 98.2 [96.6 to 99.8] | 97.1 [95.2 to 99.1]
  Week 56 | 95.3 [92.8 to 97.8] | 95.0 [92.4 to 97.5]
  Week 60 | 95.7 [93.3 to 98.1] | 96.0 [93.8 to 98.3]
  Week 64 | 98.2 [96.7 to 99.7] | 96.8 [94.7 to 98.8]
  Week 68 | 97.5 [95.6 to 99.3] | 97.5 [95.7 to 99.3]
  Week 72 | 96.4 [94.2 to 98.6] | 94.9 [92.4 to 97.5]

36. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Absence of Intraretinal Fluid and Subretinal Fluid in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 18
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 4 | 37.8 [32.1 to 43.4] | 40.8 [35.2 to 46.4]
  Week 8 | 50.9 [45.3 to 56.5] | 54.1 [48.4 to 59.9]
  Week 12 | 63.8 [58.2 to 69.4] | 56.3 [50.5 to 62.1]
  Week 16 | 67.1 [61.6 to 72.6] | 72.6 [67.4 to 77.8]
  Week 20 | 66.0 [60.5 to 71.5] | 66.0 [60.5 to 71.6]
  Week 24 | 67.4 [61.9 to 72.9] | 64.3 [58.6 to 69.9]
  Week 28 | 53.0 [47.2 to 58.7] | 46.9 [41.1 to 52.8]
  Week 32 | 67.4 [61.9 to 72.9] | 64.6 [59.0 to 70.2]
  Week 36 | 60.5 [54.8 to 66.3] | 54.2 [48.4 to 59.9]
  Week 40 | 50.4 [44.6 to 56.2] | 47.3 [41.5 to 53.2]
  Week 44 | 69.6 [64.2 to 74.9] | 63.6 [57.9 to 69.2]
  Week 48 | 74.7 [69.6 to 79.8] | 65.4 [59.8 to 70.9]
  Week 52 | 55.5 [49.6 to 61.3] | 55.6 [49.8 to 61.4]
  Week 56 | 58.0 [52.2 to 63.8] | 57.8 [52.0 to 63.6]
  Week 60 | 73.9 [68.8 to 79.1] | 70.4 [65.1 to 75.7]
  Week 64 | 75.4 [70.5 to 80.4] | 69.3 [64.0 to 74.7]
  Week 68 | 68.9 [63.4 to 74.3] | 68.3 [62.8 to 73.7]
  Week 72 | 70.7 [65.3 to 76.0] | 71.1 [65.8 to 76.4]

37. Secondary Outcome: Part 2: Change From Week 24 in BCVA in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 1
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Participants with evaluable Week 24 BCVA were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Groups:
- Arm A: Faricimab Q4W to Faricimab PTI (Part 2): In Part 2 (from Week 24 to Week 72), participants received faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure was administered during study visits at which no faricimab treatment was administered (according to the PTI dosing regimen).
- Arm B: Aflibercept Q4W to Faricimab PTI (Part 2): In Part 2 (from Week 24 to Week 72), participants received faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure was to be administered during study visits at which no faricimab treatment was administered (according to the PTI dosing regimen).
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 254 | 247
ETDRS Letters
  Week 28 | -0.3 [-0.8 to 0.3] | -0.1 [-0.6 to 0.5]
  Week 32 | 0.5 [-0.1 to 1.0] | 0.0 [-0.6 to 0.5]
  Week 36 | 0.5 [-0.2 to 1.2] | 0.6 [-0.1 to 1.2]
  Week 40 | 0.3 [-0.4 to 1.1] | 0.4 [-0.3 to 1.2]
  Week 44 | 1.1 [0.3 to 1.9] | 0.3 [-0.5 to 1.1]
  Week 48 | 1.1 [0.3 to 2.0] | 0.7 [-0.1 to 1.6]
  Week 52 | 1.1 [0.2 to 2.0] | 0.9 [0.0 to 1.8]
  Week 56 | 0.4 [-0.5 to 1.4] | 0.6 [-0.3 to 1.6]
  Week 60 | 1.0 [0.1 to 2.0] | 1.1 [0.1 to 2.0]
  Week 64 | 0.9 [0.0 to 1.9] | 1.2 [0.2 to 2.2]
  Week 68 | 1.2 [0.2 to 2.1] | 1.3 [0.4 to 2.2]
  Week 72 | 1.5 [0.5 to 2.5] | 1.3 [0.3 to 2.3]

38. Secondary Outcome: Part 2: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Week 24 in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 28 | 85.5 [81.4 to 89.6] | 84.1 [79.8 to 88.3]
  Week 32 | 89.1 [85.5 to 92.7] | 87.7 [83.9 to 91.5]
  Week 36 | 89.5 [85.9 to 93.1] | 88.4 [84.7 to 92.2]
  Week 40 | 89.5 [85.9 to 93.0] | 88.0 [84.2 to 91.8]
  Week 44 | 89.9 [86.3 to 93.4] | 86.3 [82.2 to 90.3]
  Week 48 | 89.5 [85.9 to 93.1] | 86.6 [82.6 to 90.6]
  Week 52 | 89.9 [86.3 to 93.4] | 87.7 [83.9 to 91.6]
  Week 56 | 88.0 [84.3 to 91.8] | 86.6 [82.6 to 90.6]
  Week 60 | 88.8 [85.1 to 92.5] | 87.0 [83.0 to 90.9]
  Week 64 | 89.5 [85.9 to 93.1] | 86.6 [82.6 to 90.6]
  Week 68 | 88.4 [84.7 to 92.1] | 87.0 [83.0 to 90.9]
  Week 72 | 88.4 [84.7 to 92.1] | 87.0 [83.0 to 90.9]

39. Secondary Outcome: Part 2: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Week 24 in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 28 | 84.8 [80.6 to 89.0] | 82.3 [77.8 to 86.7]
  Week 32 | 88.8 [85.1 to 92.5] | 85.9 [81.8 to 89.9]
  Week 36 | 87.3 [83.4 to 91.2] | 87.0 [83.0 to 90.9]
  Week 40 | 87.7 [83.8 to 91.5] | 86.3 [82.2 to 90.3]
  Week 44 | 88.8 [85.1 to 92.5] | 85.5 [81.4 to 89.7]
  Week 48 | 88.4 [84.7 to 92.2] | 85.2 [81.0 to 89.3]
  Week 52 | 88.4 [84.7 to 92.2] | 85.2 [81.0 to 89.3]
  Week 56 | 86.2 [82.2 to 90.2] | 83.4 [79.0 to 87.7]
  Week 60 | 86.9 [83.0 to 90.9] | 83.4 [79.0 to 87.7]
  Week 64 | 86.9 [83.0 to 90.9] | 85.2 [81.0 to 89.4]
  Week 68 | 86.6 [82.6 to 90.6] | 85.5 [81.4 to 89.7]
  Week 72 | 86.6 [82.6 to 90.6] | 85.5 [81.4 to 89.7]

40. Secondary Outcome: Part 2: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Week 24 in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 28 | 74.6 [69.5 to 79.7] | 73.6 [68.5 to 78.8]
  Week 32 | 80.0 [75.4 to 84.7] | 77.2 [72.3 to 82.1]
  Week 36 | 79.7 [75.0 to 84.4] | 79.0 [74.2 to 83.8]
  Week 40 | 78.6 [73.8 to 83.4] | 78.3 [73.5 to 83.1]
  Week 44 | 83.3 [79.0 to 87.7] | 76.9 [71.9 to 81.9]
  Week 48 | 82.6 [78.2 to 87.0] | 79.4 [74.6 to 84.1]
  Week 52 | 81.5 [77.0 to 86.0] | 79.4 [74.6 to 84.1]
  Week 56 | 76.4 [71.5 to 81.3] | 78.3 [73.5 to 83.1]
  Week 60 | 79.0 [74.2 to 83.7] | 77.2 [72.3 to 82.1]
  Week 64 | 77.9 [73.0 to 82.8] | 76.1 [71.1 to 81.1]
  Week 68 | 78.2 [73.4 to 83.1] | 76.5 [71.6 to 81.5]
  Week 72 | 77.5 [72.7 to 82.4] | 77.6 [72.7 to 82.5]

41. Secondary Outcome: Part 2: Percentage of Participants Avoiding a Loss of >0 Letters in BCVA From Week 24 in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 277
Percentage of participants
  Week 28 | 46.4 [40.6 to 52.3] | 51.3 [45.4 to 57.1]
  Week 32 | 55.4 [49.6 to 61.2] | 54.2 [48.3 to 60.0]
  Week 36 | 55.1 [49.2 to 60.9] | 52.7 [46.9 to 58.6]
  Week 40 | 56.2 [50.4 to 62.0] | 55.2 [49.4 to 61.1]
  Week 44 | 62.4 [56.7 to 68.0] | 56.0 [50.1 to 61.8]
  Week 48 | 63.8 [58.2 to 69.4] | 56.6 [50.9 to 62.4]
  Week 52 | 59.8 [54.1 to 65.5] | 58.5 [52.7 to 64.3]
  Week 56 | 57.2 [51.5 to 63.0] | 57.4 [51.5 to 63.2]
  Week 60 | 58.0 [52.1 to 63.8] | 60.3 [54.5 to 66.0]
  Week 64 | 62.0 [56.3 to 67.7] | 56.6 [50.8 to 62.5]
  Week 68 | 60.9 [55.1 to 66.6] | 58.8 [53.1 to 64.6]
  Week 72 | 63.0 [57.4 to 68.7] | 58.1 [52.3 to 63.9]

42. Secondary Outcome: Part 2: Percentage of Participants on Different Treatment Intervals at Week 68
Description: In Part 2 of the study, participants in both the faricimab Q4W and aflibercept Q4W arms in Part 1 received 6 mg faricimab intravitreal injections administered according to a personalized treatment interval (PTI) dosing regimen in intervals between Q4W and Q16W. At faricimab dosing visits, treatment intervals were maintained or adjusted (i.e., increased by 4 weeks or decreased by 4, 8, or 12 weeks), based on central subfield thickness (CST) and BCVA values.
Time Frame: Week 68
Population: The analysis population included all randomized participants who had not discontinued the study at Week 68.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 248 | 244
Percentage of participants
  Once Every 4 Weeks (Q4W) | 22.6 [17.4 to 27.8] | 25.0 [19.6 to 30.4]
  Once Every 8 Weeks (Q8W) | 13.3 [9.1 to 17.5] | 18.0 [13.2 to 22.9]
  Once Every 12 Weeks (Q12W) | 11.7 [7.7 to 15.7] | 9.4 [5.8 to 13.1]
  Once Every 16 Weeks (Q16W) | 52.4 [46.2 to 58.6] | 47.5 [41.3 to 53.8]

43. Secondary Outcome: Part 2: Number of Study Drug Injections Received in the Study Eye From Week 24 Through Week 72
Time Frame: From Week 24 to Week 72
Population: Safety-Evaluable Population: All participants randomized in the study who received at least one injection of active study drug in the study eye. For Part 2, the safety analysis included: in Arm A, all participants with Week 24 treatment or dose hold, or if none, follow-up beyond Day 168; in Arm B, all participants who received at least one faricimab dose.
Measure: Median (Full Range); unit: Injections
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 270 | 267
Injections | 4.0 [1 to 12] | 4.0 [1 to 12]

44. Secondary Outcome: Incidence and Severity of Ocular Adverse Events in the Study Eye, With Severity Determined According to Adverse Event Severity Grading Scale
Description: This analysis of adverse events (AEs) only includes ocular AEs that occurred in the study eye. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. Ocular AEs of special interest included the following: Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation (IOI).
Time Frame: Part 1: From first dose up to Week 24; Part 2: from Week 24 through Week 72
Population: Safety-Evaluable Population: All participants randomized in the study who received at least one injection of active study drug (faricimab or aflibercept) in the study eye. For Part 2, the safety analysis included: in Arm A, all participants with Week 24 treatment or dose hold, or if none, follow-up beyond Day 168 (6 were excluded); in Arm B, all participants who received at least one faricimab dose (7 were excluded).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 274 | 270 | 267
Participants
  Adverse Event (AE) | 45 | 56 | 76 | 81
  AE by Severity: Mild | 40 | 47 | 50 | 64
  AE by Severity: Moderate | 4 | 8 | 25 | 16
  AE by Severity: Severe | 0 | 1 | 1 | 1
  AE by Severity: Missing | 1 | 0 | 0 | 0
  Serious Adverse Event (SAE) | 3 | 2 | 4 | 3
  AE Leading to Withdrawal from Study Treatment | 0 | 0 | 0 | 1
  Treatment Related AEs | 1 | 3 | 7 | 8
  Treatment Related SAEs | 0 | 0 | 0 | 0
  Any AE of Special Interest (AESI) | 1 | 2 | 1 | 1
  AESI: Drop in Visual Acuity Score ≥30 | 1 | 2 | 1 | 1

45. Secondary Outcome: Incidence of Ocular Adverse Events in the Fellow Eye
Description: This analysis of adverse events (AEs) only includes ocular AEs that occurred in the fellow eye. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. Ocular AEs of special interest included the following: Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation (IOI).
Time Frame: Part 1: From first dose up to Week 24; Part 2: from Week 24 through Week 72
Population: Safety-Evaluable Population: All participants randomized in the study who received at least one injection of active study drug (faricimab or aflibercept) in the study eye. For Part 2, the safety analysis included: in Arm A, all participants with Week 24 treatment or dose hold, or if none, follow-up beyond Day 168 (6 excluded); in Arm B, all participants who received at least one faricimab dose (7 excluded).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 274 | 270 | 267
Participants
  Adverse Event (AE) | 25 | 21 | 37 | 30
  Serious Adverse Event (SAE) | 0 | 0 | 0 | 0
  Any AE of Special Interest (AESI) | 0 | 0 | 0 | 0

46. Secondary Outcome: Incidence of Non-Ocular Adverse Events
Description: This analysis of adverse events (AEs) only includes non-ocular (systemic) AEs. Investigators sought information on adverse events (AEs) at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. The non-ocular AE of special interest was: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: Part 1: From first dose up to Week 24; Part 2: from Week 24 through Week 72
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 274 | 270 | 267
Participants
  Adverse Event (AE) | 94 | 99 | 136 | 126
  Serious Adverse Event (SAE) | 9 | 16 | 25 | 23
  AE Leading to Withdrawal from Study Treatment | 1 | 0 | 0 | 3
  Any AE of Special Interest (AESI) | 0 | 0 | 0 | 0

47. Secondary Outcome: Plasma Concentration of Faricimab Over Time
Time Frame: Predose at Day 1 (Baseline), Weeks 4, 24, 28, 52, and 72
Population: Pharmacokinetic-Evaluable Population: All safety- evaluable participants randomized to faricimab arm or who received faricimab with at least one plasma sample, provided sufficient dosing information (dose and dosing time) is available. The number analyzed indicates all participants who provided a PK sample at a given timepoint.
Measure: Mean (Standard Deviation); unit: microgram per millilitre (μg/mL)
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 276 | 268
microgram per millilitre (μg/mL)
  Baseline: number analyzed (Participants) | 273 | 0
  Baseline | 0.0000 (0.0000) |
  Week 4: number analyzed (Participants) | 264 | 0
  Week 4 | 0.0215 (0.0160) |
  Week 24: number analyzed (Participants) | 247 | 241
  Week 24 | 0.0220 (0.0181) | 0.0005 (0.0006)
  Week 28: number analyzed (Participants) | 238 | 242
  Week 28 | 0.0040 (0.0072) | 0.0025 (0.077)
  Week 52: number analyzed (Participants) | 231 | 224
  Week 52 | 0.0061 (0.0110) | 0.0097 (0.0156)
  Week 72: number analyzed (Participants) | 231 | 229
  Week 72 | 0.0076 (0.0109) | 0.0087 (0.0146)

48. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Faricimab at Baseline and Post-Baseline During the Study
Description: Anti-drug antibodies (ADAs) against fariciamb were detected in plasma using a validated bridging enzyme-linked immunosorbent assay (ELISA). The number of participants with treatment-emergent ADA-positive samples includes post-baseline evaluable participants with at least one treatment-induced (defined as having an ADA-negative sample or missing sample at baseline and any positive post-baseline sample) or treatment-boosted (defined as having an ADA-positive sample at baseline and any positive post-baseline sample with a titer that is equal to or greater than 4-fold baseline titer) ADA-positive sample during the study treatment period. Treatment-unaffected ADA-positive is a post-baseline sample with a titer that is lower than 4-fold the ADA-positive baseline titer (faricimab arm) or the ADA-positive titer prior to first faricimab injection (aflibercept arm).
Time Frame: Predose at Day 1 (Baseline), Weeks 4, 24, 28, 52, and 72
Population: The immunogenicity analysis included all participants with an evaluable ADA sample. At baseline, evaluable participants were those with an ADA sample prior to faricimab injection, including those who did not receive study treatment; post-baseline, evaluable participants were those with an ADA sample after having received at least one dose of faricimab.
Measure: Count of Participants; unit: Participants
Groups:
- All Faricimab Participants: This immunogenicity analysis group represents all participants with an evaluable ADA sample. At baseline, evaluable participants were those with an ADA sample prior to faricimab injection, including those who did not receive study treatment; post-baseline, evaluable participants were those with an ADA sample after having received at least one dose of faricimab.
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2) | All Faricimab Participants
Number analyzed (Participants) | 274 | 266 | 540
Participants
  Baseline (BL): Total ADA-Positive | 3 | 4 | 7
  Post-BL: Total ADA-Positive: number analyzed (Participants) | 274 | 264 | 538
  Post-BL: Total ADA-Positive | 33 | 23 | 56
  Post-BL: Treatment-Emergent ADA-Positive: number analyzed (Participants) | 274 | 264 | 538
  Post-BL: Treatment-Emergent ADA-Positive | 32 | 21 | 53
  Post-BL: Treatment-Unaffected ADA-Positive: number analyzed (Participants) | 274 | 264 | 538
  Post-BL: Treatment-Unaffected ADA-Positive | 1 | 2 | 3

ADVERSE EVENTS:
Time Frame: Part 1: From first dose up to Week 24; Part 2: from Week 24 through Week 72
Description: Adverse events (AEs) are reported for the safety population, which includes all participants who received ≥1 injection of active study drug (faricimab or aflibercept) in the study eye. For Part 2, safety analysis included: in Arm A, those with Week 24 treatment or dose hold, or if none, follow-up beyond Day 168; in Arm B, those who received ≥1 faricimab dose. For ocular AEs, the number of participants and events reported per term are specified to have occurred in the study eye or the fellow eye.
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
All-Cause Mortality (participants affected / at risk) | 1/276 | 0/274 | 1/270 | 2/267
Serious Adverse Events (participants affected / at risk) | 12/276 | 17/274 | 29/270 | 26/267
Other Adverse Events (participants affected / at risk) | 62/276 | 69/274 | 92/270 | 87/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Faricimab Q4W (Part 1) (N=276) | Arm B: Aflibercept Q4W (Part 1) (N=274) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) (N=270) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2) (N=267)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Retinal ischaemia (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) — AEs occurred in the study eye
Retinal vein occlusion (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — AEs occurred in the study eye
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — AEs occurred in the study eye
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urogenital prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertebral artery hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — AEs occurred in the study eye
Macular ischaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Retinal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Tractional retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Faricimab Q4W (Part 1) (N=276) | Arm B: Aflibercept Q4W (Part 1) (N=274) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) (N=270) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2) (N=267)
COVID-19 (Infections and infestations) | 10 (10) | 16 (16) | 32 (32) | 25 (25)
Hypertension (Vascular disorders) | 20 (21) | 7 (7) | 14 (14) | 8 (8)
Conjunctival haemorrhage (Eye disorders) | 8 (9) | 10 (11) | 11 (11) | 10 (11) — AEs occurred in the study eye
Dry eye (Eye disorders) | 5 (5) | 9 (9) | 4 (5) | 4 (4) — AEs occurred in the study eye
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 10 (10) | 5 (6) | 4 (4)
Nasopharyngitis (Infections and infestations) | 6 (6) | 6 (6) | 7 (8) | 10 (12)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5) | 6 (8) | 9 (11)
Cataract (Eye disorders) | 2 (2) | 1 (1) | 9 (9) | 9 (9) — AEs occurred in the study eye
Vitreous detachment (Eye disorders) | 4 (4) | 2 (2) | 7 (7) | 9 (9) — AEs occurred in the study eye
Retinal vein occlusion (Eye disorders) | 0 (0) | 2 (3) | 9 (12) | 8 (10) — AEs occurred in the study eye
Intraocular pressure increased (Investigations) | 1 (2) | 8 (8) | 13 (21) | 8 (11) — AEs occurred in the study eye
Vitreous floaters (Eye disorders) | 7 (7) | 6 (6) | 0 (0) | 9 (9) — AEs occurred in the study eye
Macular oedema (Eye disorders) | 1 (1) | 2 (2) | 10 (11) | 5 (8) — AEs occurred in the study eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT04740905/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT04740905/SAP_001.pdf